CLINICAL TRIAL: NCT02901184
Title: Spironolactone Initiation Registry Randomized Interventional Trial in Heart Failure With Preserved Ejection Fraction, SPIRRIT-HFPEF
Brief Title: Spironolactone Initiation Registry Randomized Interventional Trial in Heart Failure With Preserved Ejection Fraction
Acronym: SPIRRIT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Karolinska University (Other); Duke Clinical Research Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-2015-030; U01HL134679-01 (NIH); U01HL134694-02 (NIH)
Record Dates: First submitted 2016-09-09; First posted 2016-09-15 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Spironolactone; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spironolactone treatment (Active Comparator): Spironolactone will be prescribed by the Investigator and filled by patient at conventional pharmacies as 25 mg tablets. The treatment will be on top of standard care. Initial dose is 25 mg/day, which will be increased to target dose 50 mg/day if tolerated. Eplerenone can be prescribed if spironolactone is not tolerated.
  Interventions: Drug: Spironolactone
- Standard care alone (Placebo Comparator): Patients in the control arm will get the standard care alone
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Spironolactone — Treatment with Spironolactone tablets on top of standard care
  Arms: Spironolactone treatment
Other: Standard care — Standard care does not involve Spironolactone
  Arms: Standard care alone

SUMMARY:
Heart failure with preserved ejection fraction (HFPEF) is common and deadly but without therapy. Inconclusive studies such as TOPCAT (Treatment of Preserved Cardiac Function Heart Failure With an Aldosterone Antagonist) suggest spironolactone may be effective in HFPEF, but it is generic and will not be studied by industry.

SPIRRIT is a unique Registry-Randomized Clinical Trial (RRCT) that will test the hypothesis that spironolactone plus standard of care compared to standard of care alone reduces the composite of CV mortality and HF hospitalization as follows:

Population: HFPEF patients in the Swedish Heart Failure Registry and HFPEF patients in US. HFPEF defined as symptoms/signs of HF, elevated NTproBNP (B-type Natriuretic Peptide; N-terminal pro b-type Natriuretic Peptide) and EF>=40%. Intervention and control: Randomized 1:1 to intervention: spironolactone + usual care vs. control: usual care alone.

Outcome: Primary outcome cardiovascular death or time to HF hospitalization. Secondary outcomes include hospitalization for various causes, adverse events and treatment adherence. In Sweden outcomes are obtained automatically by linking with the Population, Patient and Drug Dispensed Registries. In the US, outcomes will be reported by sites and supplemented by data from a call center. The trial is event-driven with enrollment 7 years and study duration 9 years. For the primary outcome (CV Death or first HF hospitalization) with an event target of 721 events the sample size requires 1985 patients conservatively rounded to approximately 2000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥50 years
* Stable heart failure defined by symptoms and signs of heart failure as judged by local Investigator
* Left ventricular ejection fraction (LVEF) ≥40% recorded in last 12 months (stratified to max 2/3rd in either 40-49% or ≥50% group)
* Elevated natriuretic peptide levels, as defined by any of the following:

  1. most recent NT-proBNP >300 ng/L (or BNP>100 pg/mL) in sinus rhythm at time of blood sampling; adjustments may be made for BMI according to table 3.
  2. most recent NT-proBNP >750 ng/L (or BNP >250 pg/mL) in atrial fibrillation at time of blood sampling; adjustments may be made for BMI according to table 3.
  3. NT-proBNP >1200 ng/L (or BNP >400 pg/mL) within the last 12 months even if most recent value is lower.
* Regular use of loop diuretics, defined as daily or most days of the week
* NYHA Class II-IV

Exclusion Criteria:

Previously enrolled in this study

* Known Ejection Fraction < 40% ever
* Current absolute indication or contraindication for MRA (mineral receptor antagonist) in judgement of Investigator
* Known chronic liver disease
* Probable alternative explanations for symptoms:

  * Known primary cardiomyopathy (hypertrophic, constrictive, restrictive, infiltrative, congenital)
  * Primary hemodynamically significant valve disease
  * Right-sided HF not due to left-sided HF
  * Significant chronic pulmonary disease defined by Investigator or by requirement for home O2
  * Symptomatic anemia, defined as Hemoglobin < 10 g/dL (100 g/L )
* Heart transplant or LVAD (left ventricular assist device) recipient
* Presence of cardiac resynchronization therapy (CRT) device
* Systolic blood pressure <90 or >160 mmHg
* K (potassium) >5.0 mmol/L
* eGFR (estimated glomerular filtration rate) by MDRD (Modification of Diet in Renal Disease) < 30 ml/min/1.73m2 or creatinine > 2.5 mg/dL (221 µmol/L )
* Current lithium use
* Current dialysis
* Actual or potential for pregnancy
* Participation in another interventional clinical trial where a mineralocorticoid receptor antagonist is studied
* Any condition that in the opinion of the Investigator may interfere with adherence to trial protocol

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate for total heart failure (HF) hospitalizations or cardiovascular (CV) death | Collected at data base lock, five (5) years after study start (US: continuously until 5 years after study start)
  Sweden: Information on Death from the Swedish Causes of death registry and information on hospitalization collected from Swedish Patient Registry US: Collected in eCRF or via call center interview

SECONDARY OUTCOMES:
Time to CV Death or first HF hospitalization | Collected at data base lock, five (5) years after study start (US: continuously until 5 years after study start)
  Sweden: Information on Death from the Swedish Causes of death registry US: Collected in eCRF or via call center interview
Time to CV Death | Collected at data base lock, five (5) years after study start (US: continuously until 5 years after study start)
  Sweden: Information on Death from the Swedish Causes of death registry US: Collected in eCRF or via call center interview
Incidence rate for total HF hospitalizations | Collected at data base lock, five (5) years after study start (US: continuously until 5 years after study start)
  Sweden: Information on Death from the Swedish Causes of death registry and information on hospitalization collected from Swedish Patient Registry.
  US: Collected in eCRF or via call center interview
Time to HF hospitalizations | Collected at data base lock, five (5) years after study start (US: continuously until 5 years after study start)
  Sweden: Information on information on hospitalization collected from Swedish Patient Registry.
  US: Collected in eCRF or via call center interview
Time to all-cause mortality | Collected at data base lock, five (5) years after study start
  Sweden: Information on Death from the Swedish Causes of death registry. US: Collected in eCRF or via call center interview
Incidence rate for all-cause hospitalizations | Collected at data base lock, five (5) years after study start (US: continuously until 5 years after study start)
  Sweden: Information on information on hospitalization collected from Swedish Patient Registry.
  US: Collected in eCRF or via call center interview
Time to all-cause hospitalizations | Collected at data base lock, five (5) years after study start (US: continuously until 5 years after study start)
  Sweden: Information on information on hospitalization collected from Swedish Patient Registry.
  US: Collected in eCRF or via call center interview
Incidence rate for all-cause hospitalizations or all-cause mortality | Collected at data base lock, five (5) years after study start (US: continuously until 5 years after study start)
  Sweden: Information on Death from the Swedish Causes of death registry and information on hospitalization collected from Swedish Patient Registry.
  US: Collected in eCRF or via call center interview

CONTACTS AND LOCATIONS:
Overall Officials: Lars H Lund, MD, PhD, Principal Investigator — Karolinska Institutet; Bertram Pitt, Principal Investigator — University of Michigan
Locations (78):
- United States (38):
  - Advanced Cardiovascular LLC, Alexander City, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner - University Medical Group, Tucson, Arizona
  - MedStar Cardiovascular Research Network, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Wellstar Health System, Inc., Marietta, Georgia
  - Queens Medical Center, Honolulu, Hawaii
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Shady Grove Adventist Hospital, Rockville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Charles River Medical Associates, Natick, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Ascension Genesys Hospital, Grand Blanc, Michigan
  - The Heart House Haddon Heights, Haddon Heights, New Jersey
  - Rutgers University - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - University at Buffalo, Buffalo, New York
  - Northwell Health - Manhasset, Manhasset, New York
  - Mount Sinai Medical Cente, New York, New York
  - Mid Carolina Cardiology Research, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Stern Cardiovascular Center, Germantown, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Miami Hospital, Miami, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Sweden (40):
  - Angereds närsjukhus, Angered
  - Hälsostaden Ängelholms sjukhus, Ängelholm
  - Falu lasarett, Falun
  - Närsjukvården i Finspång, Finspång
  - Vårdcentralen Centrum i Flen, Flen
  - Sahgrenska University Hospital Östra, Gothenburg
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Hemse Vårdcentral, Hemse
  - Karolinska University Hospital, Huddinge
  - Länssjukhuset Ryhov, Jönköping
  - Blekingesjukhuset, Karlskrona
  - Hjärtmottagningen, Centralsjukhuset, Karlstad
  - Västmanlands sjukhus Köping, Köping
  - Centralsjukhuset Kristianstad, Kristianstad
  - Lasarettet i Landskrona, Landskrona
  - Skaraborgs sjukhus i Lidköping, Lidköping
  - Linköpings Universitetssjukhus, Linköping
  - VO Akut- och internmedicin, Skånes Universitetssjukhus, Lund
  - Capio Citykliniken, Lund
  - FO Kranskärl/Svikt, Skånes Universitetssjukhus, Lund
  - Hjärtavdelningen, Skånes Universitetssjukhus, Malmo
  - Kliniska forskningsenheten Skånes Universitetssjukhus, Malmo
  - Mariefreds Vårdcentral, Mariefred
  - Sahlgrenska University Hospital Mölndal, Mölndal
  - Kardiologikliniken, Vrinnevisjukhuset, Norrköping
  - Oskarshamns sjukhus, Oskarshamn
  - Örebro University Hospital, Örebro
  - Skellefteå lasarett, Skellefteå
  - Karolinska University Hospital, Solna
  - Södertälje sjukhus, Södertälje
  - VO Kardiologi, Södersjukhuset AB, Stockholm
  - Capio S:t Görans sjukhus AB, Stockholm
  - Danderyds sjukhus AB, Stockholm
  - Länssjukhuset Sundsvall-Härnösand, Sundsvall
  - Sundsvalls Vårdcentral, Sundsvall
  - Uppsala University Hospital, Cardiology dept, Uppsala
  - Uppsala University Hospital, Internal Medicine dept, Uppsala
  - Medicinkliniken, Hallands sjukhus, Varberg
  - Västmanlands sjukhus Västerås, Västerås
  - Västerviks sjukhus, Västervik

IPD SHARING:
Plan to Share IPD: Yes